CLINICAL TRIAL: NCT04916223
Title: Study to Determine Therapeutic Massage Dosing to Improve Quality of Life in Hospitalized Patients Receiving Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-260
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Cancer; Heart Failure; COPD; Sepsis; HIV Infections; ESRD; Trauma; Stroke
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive; Sepsis; HIV Infections; Kidney Failure, Chronic; Wounds and Injuries; Stroke | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 x 10-minute massage (Experimental): Subject receives a 10-minute massage daily for three consecutive days
  Interventions: Other: Therapeutic massage
- 3 x 20-minute massage (Experimental): Subject receives a 20-minute massage daily for three consecutive days
  Interventions: Other: Therapeutic massage
- Single 20-minute massage (Active Comparator): Subject receives one 20-minute massage
  Interventions: Other: Therapeutic massage

INTERVENTIONS:
Other: Therapeutic massage — The massage therapists were scheduled on a rotating schedule with two alternates scheduled for each day to ensure adherence to assigned study arm and to avoid "therapist effect" as much as possible. For each enrolled subject, the therapist assessed the subject and created a treatment plan depending on his/her individual needs and preferences. For example, if a subject reported bothersome lower extremity pain, the therapist might focus the massage on that lower extremity or might avoid massaging that lower extremity, depending solely on the preference of the subject. Massage duration was determined by the assigned study arm.

SUMMARY:
Therapeutic massage is the most common non-traditional treatment option offered to improve quality of life, provide comfort and decrease pain in hospice and palliative care settings outside the hospital. Three systematic reviews of data in general pain, surgical and cancer populations found massage to be effective for treating pain versus active comparators.

Given the remarkable negative impact on QOL experienced by patients hospitalized with a serious progressive illness, a nationwide opioid crisis in the setting of public concern for untreated pain, and patient demand for integrative therapies, we wish to investigate non-traditional methods of supporting patients in pain and providing clinicians with viable alternatives. Unfortunately, very little is known about optimal delivery of massage interventions in the hospital setting, including dosing parameters such as time and frequency

We conducted a single center comparative effectiveness study to evaluate therapeutic massage "dosing" to improve self-reported quality-of-life in hospitalized patients receiving palliative care consultation.

DETAILED DESCRIPTION:
Palliative care (PC) provides expert symptom management and communication skills for patients and families facing serious life-limiting illness in the hospital. Many such patients experience lower quality of life (QOL) due to moderate-severe pain or other symptoms and require strong pharmacotherapies - often controlled substances such as opioids or benzodiazepines - to alleviate associated distress. A major tenet of quality supportive care is the combination of many types of therapy, both pharmacologic and nonpharmacologic. Patients with serious life-limiting illnesses often rely on the use of nonpharmacologic therapies to manage pain or other symptoms at home. However, implementing complementary therapies in the hospital setting can be challenging and thus they are rarely available for hospitalized patients with serious illness. Patients often request non-drug options, but medications remain the mainstay of treating pain while hospitalized.

Therapeutic massage is the most common non-traditional treatment option offered to improve quality of life, provide comfort and decrease pain in hospice and palliative care settings outside the hospital. Nevertheless, there remains limited data describing the impact of therapeutic massage in hospitalized patients receiving palliative care.

Additionally, in the hospital setting, the logistical challenges of providing massage therapy include a number of setting-specific factors. A massage therapy session may be interrupted by care being provided by other members of the team, by personal visitors, or by the activities of his/her roommate in a semi-private room. Also, the availability of massage therapy may be such that a patient's session time is limited because of the high demand on the short amount of time a non-integrated, contracted massage therapist has to see multiple patients. Given the remarkable negative impact on QOL experienced by patients hospitalized with a serious progressive illness, a nationwide opioid crisis in the setting of public concern for untreated pain, and patient demand for integrative therapies, we wish to investigate non-traditional methods of supporting patients in pain and providing clinicians with viable alternatives. Unfortunately, very little is known about optimal delivery of massage interventions in the hospital setting, including dosing parameters such as time and frequency.

The purpose of this study is to examine the impact of different massage dosing strategies on QOL, symptom management, and satisfaction in hospitalized patients already receiving PC consultation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* hospitalized, receiving inpatient palliative care consultation for any indication

Exclusion Criteria:

* unable to complete surveys in English
* on negative-pressure isolation
* unstable spine
* platelets < 10,000
* received massage in last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post-intervention in McGill Quality of Life Questionnaire Single Item | Baseline and one day post intervention
  The McGill QOL Questionnaire is a validated reliable tool to evaluate self-reported QOL. One item in the Questionnaire has been shown to effectively assess subject's self-reported QOL.

SECONDARY OUTCOMES:
Change from baseline to post-intervention in Edmonton Symptom Assessment Scale | Baseline and one day post intervention
  The Edmonton Symptom Assessment Scale is a validated, reliable instrument developed to measure 9 different common symptoms in advanced illness
Change from baseline to post-intervention in National Comprehensive Cancer Network Distress Thermometer | Baseline and one day post intervention
  The NCCN Distress Thermometer is an 11-point Likert scale tool to self-report general distress between 0 (no distress) and 10 (extreme distress)
Change from baseline to post-intervention in Peace Questionnaire | Baseline and one day post intervention
  We adapted a single-item probe of spiritual concerns ("are you at peace?") to a 5-point Likert scale to self-report experience of being at peace, where 0=experiencing no peace and 5=experiencing total peace.
Satisfaction with assigned intervention | One day post intervention
  We developed a post-intervention Patient Satisfaction Survey that included pain-related questions from the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey, modified to reference the current hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No